CLINICAL TRIAL: NCT03351660
Title: Diagnostic Value of the CardioSecur Connected EcG in General Care: The Connected EGG-study.
Brief Title: CardioSecur Connected Electrocardiography in General Care
Acronym: CARDIOSECUR
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RCP-0063
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Heart Diseases; Connected ECG; Family Practice
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: connected ECG — Cardiosecur allows the realization of a 15 or 22 leads ECG with only 4 electrodes connected to a tablet with an automatic interpretation function

SUMMARY:
Heart disease symptoms are a frequent reason of consultation in general medical practice. Only a few general practitioners are equipped with a 12 lead Electrocardiography (ECG) whereas this test is extremely useful for diagnosis orientation in cases of cardiac diseases.Cardiosecur allows the realization of a 15 or 22 leads ECG with only 4 electrodes connected to a smartphone or a tablet with an automatic interpretation function. The goal of the study is to evaluate the diagnostic value of Cardiosecur device regarding cardiac symptoms in family practice.

DETAILED DESCRIPTION:
This study will be a multicenter, single arm, non randomized trial testing the incremental diagnosis value of Cardiosecur ECG regarding cardiac disease in general care.

Ten general practitioners will be given a Cardiosecure ACTIVE device with a tablet and perform an EKG to their consecutive patients who meet the inclusion criteria.

Inclusion criteria

* Recent cardiovascular symptom < 7 days (chest pain, dyspnea, palpitation, heart failure or transient loss of consciousness) or physical examination leading in possible cardiac cause.
* Aged over 18 years
* signed the informed consent

  * A questionnaire regarding the diagnosis orientation based on the patients' symptoms and physical examination will be given to GPs before and after the ECG realization and automatic interpretation to evaluate whether the ECG modified the diagnosis.

If the GP need further exploration to conclude or if the patient is oriented to an hospital or a specialist, the reference diagnosis will be defined at the end of these explorations. Otherwise, the diagnostic will be defined at the end of the GP consultation.

* A questionnaire regarding the ease of use of the Cardiosecure device will be filled by the patients.
* Time for ECG realization will be recorded.
* All the ECG and their automatic interpretation will be stored anonymously according to bioethics laws and then reviewed by 2 experienced cardiologists blinded to the results of the automatic interpretation. The interobserver reproducibility as well as the comparison with the Cardiosecur automatic interpretation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Recent cardiovascular symptoms < 7 days (chest pain, dyspnea, palpitations, heart failure or transient loss of consciousness) or physical examination suggesting cardiac disease.
* Patients aged over 18 years
* Signed the informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients consulting a family doctor and presenting clinical manifestions of heart disease
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Performance of ECG Cardiosecur | Baseline
  Proportion of correct diagnosis before and after Cardiosecur

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric Menet, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (9):
- France (9):
  - Aire-sur-la-Lys
  - Chenôve
  - Cysoing
  - Dijon
  - Iteuil
  - Montreuil-sur-Mer
  - Poitiers
  - Roubaix
  - Vervins

IPD SHARING:
Plan to Share IPD: No